CLINICAL TRIAL: NCT06345911
Title: The Effectiveness of Using Animal-Themed Vacutainers to Reduce Fear and Anxiety in Children During Bloodletting
Brief Title: Do Vacutainers With Animal Characters Reduce Fear and Anxiety?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Burdur Mehmet Akif Ersoy University (Other)
Responsible Party: Principal Investigator, Selda Ateş Beşirik, Principal Investigator, Burdur Mehmet Akif Ersoy University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: NEU-49/899
Record Dates: First submitted 2024-03-28; First posted 2024-04-03 (Actual); Last update posted 2024-04-03 (Actual); Status verified 2024-03

CONDITIONS: Procedural Pain; Acute Pain; Fear; Anxiety
Keywords: Bloodletting; Animal Vacutainer; Procedural Pain; Fear; Distraction
MeSH Terms: conditions — Pain, Procedural; Acute Pain; Anxiety Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): The animal characters were shown to the child before the bloodletting procedure. The child was asked to choose one of them and the one chosen by the child was attached to the vacutainer.
  Interventions: Behavioral: Experimental group
- Control group (No Intervention): The child was subjected to routine bloodletting intervention with the vacutainer.

INTERVENTIONS:
Behavioral: Experimental group — The animal characters were shown to the child before the bloodletting procedure. The child was asked to choose one of them and the one chosen by the child was attached to the vacutainer. The child and their parents were taken to the blood collection room. During the bloodletting procedure, the child was asked to focus on the animal character they had chosen.
  Arms: Experimental group

SUMMARY:
The study was designed as a randomized controlled experimental research with the purpose of determining the effect of distraction by using vacutainers of three different animal characters.

DETAILED DESCRIPTION:
In the literature, it is stated that nurses should use pharmacological and non-pharmacological methods in pain and anxiety management in painful procedures. Evidence-based studies are needed to show the effectiveness of non-pharmacological methods in reducing pain during invasive procedures and to investigate the effects of easy-to-apply methods on pain. In light of this information, this study aimed to compare the effects of vacutainers of three different animal characters on fear, anxiety, and pain in children during bloodletting.

The study is a prospective, randomized and controlled trial.Children aged 4 to 7 years who required blood draw were divided into three groups; two groups: experimental and control groups. Animal characters (butterfly, peacock and rabbit) chosen by children in the experimental group was attached to the vacutainer, and then their blood was drawn. The data were obtained by face-to-face interviews with the child, parent and observer before and after the procedure. Children's pain and fear/anxiety levels were evaluated using the Children's Fear Scale and theWong-Baker FACES Pain Scale, respectively.

The study population consisted of children aged 4 to 7 years who presented to the children's blood draw room of the hospital.

Sample of the study consisted of a total of 1800 children who met the sample selection criteria and were selected via randomization method.

Data were collected using the Interview and Observation Form, Children's Fear Scale, and Wong-Baker FACES Pain Rating Scale.

ELIGIBILITY:
Inclusion Criteria:

* The child was selected by simple randomization.
* The child was between 4-7 years old.
* The child and parent were informed and their written consent was obtained prior to the procedure.
* The bloodletting procedure was performed by the same nurse.
* The child was given standard information before the bloodletting procedure.
* The needle used for the bloodletting procedure was of the same thickness.
* The child could evaluate the pain and fear scales.

Exclusion Criteria:

* The child was excluded from the study if they had the following criteria;
* The child had infection, skin integrity disturbance, and rash in the area where the procedure would be performed.
* The child had nerve damage in the previously treated area.
* The child's health status was critical and unstable.
* The child had developmental retardation that prevents them from responding to pain and fear scales.
* The child had taken any analgesic in the last 6 hours before the bloodletting procedure.
* The child did not want to participate.
* The child did not meet the selection criteria for the experimental and control groups.

Ages: 4 Years to 7 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 180 (Actual)
Dates: Start 2021-12-01 (Actual); Primary Completion 2022-02-25 (Actual); Study Completion 2022-03-30 (Actual)

PRIMARY OUTCOMES:
Children's Fear Scale | Through painful procedure completion, an average of 10 minutes
  CFS is used for measuring the child's anxiety level. CFS is a scale which makes an evaluation from 0 to 4 consisting of five facial expressions drawn to show expressions that vary from neutral expression (0=no anxiety) to scared face (4=severe anxiety).
Wong-Baker FACES Pain Rating Scale | Through painful procedure completion, an average of 10 minutes.
  In the study, pain level evaluations, the children's self-evaluations, parents' evaluations and the researcher's evaluations were carried out using the WB-FACES scale. This scale was developed by Donna Wong and Connie Morain Baker in 1988. The scale is graded between 0-10 points. A smiling face on the far left symbolizes "no pain" (0 very happy/no pain) and the pain increases from left to right. On the other hand, a crying face on the far right symbolizes "unbearable pain" (10 'hurts worst'). As the numbers increase in this scoring system, facial expressions also change referring to an increase in pain levels.

CONTACTS AND LOCATIONS:
Overall Officials: Selda Ateş Beşirik, PhD., Principal Investigator — Burdur Mehmet Akif Ersoy University
Locations (1):
- Karaman Education and Research Hospital, Karaman, Turkey (Türkiye)